CLINICAL TRIAL: NCT03743519
Title: The Efficacy of a Tart Cherry Drink for Patellofemoral Pain.
Brief Title: The Efficacy of a Tart Cherry Drink for the Treatment of Patellofemoral Pain in Recreational Athletes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Senior Lecturer, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cherry juice
Record Dates: First submitted 2018-11-10; First posted 2018-11-16 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2019-05

CONDITIONS: Patellofemoral Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Cherry juice (Experimental)
  Interventions: Dietary Supplement: Cherry juice

INTERVENTIONS:
Dietary Supplement: Cherry juice — 30 mL of tart cherry juice concentrate, which will be diluted with 200 mL of water.
  Arms: Cherry juice
Dietary Supplement: Placebo — Identical in taste and colour to the Cherry juice, but with no anthocyanin content
  Arms: Placebo

SUMMARY:
Patellofemoral pain (PFP) is the most common chronic pathology in sports medicine and physiotherapy clinics. As pain and inflammation are the main symptoms of PFP, non-steroidal anti-inflammatory and analgesic medications are often utilized to decrease pain and inflammation; however alternative treatments are increasingly being sought due to the cardiovascular and gastrointestinal side effects of traditional pain medications. Most researchers advocate conservative treatment, though there is still insufficient clarity regarding the effectiveness of conservative treatment modalities. Dietary interventions for PFP have not received any attention in clinical literature, yet there is a growing body of evidence indicating that cherries have significant anti-inflammatory, antioxidant and pain-mediating effects.

Therefore, the primary purpose of the proposed investigation was to test (using a randomized control investigation) the ability of a tart cherry juice blend to provide symptom relief in recreational athletes with PFP and to understand the biological and mechanical mechanisms behind any changes in PFP symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active
* Suffering from mild to moderate patellofemoral pain with no evidence of any other condition.

Exclusion Criteria:

* Rheumatoid arthritis or other systemic inflammatory condition
* Chronic pain syndrome
* Corticosteroid medication in last 2 months (intra-articular or oral)
* Intra-articular injections of hyaluronic acid in the last 9 months
* Pregnancy
* Diabetes
* Food allergies to cherries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) - patellofemoral scale | 6-weeks
  This is a questionnaire based measurement that allows participants to subjectively rate the extent of their patellofemoral pain symptoms. This measurement is scored on a 0-100 scale with 100 indicating no pain.

SECONDARY OUTCOMES:
COOP-WONCA - psychological wellbeing | 6-weeks
  This is a questionnaire based measurement that allows participants to subjectively rate their psychological wellbeing. This measurement provides a value that is an average score of 6 questions (overall health, daily activities, physical fitness, feelings, social activities and change in health) that range from 1-5. A lower score indicates better psychological wellbeing.
Plasma urate | 6-weeks
Creatinine | 6-weeks
human TNF-alpha | 6-weeks
High sensitivity C-reactive protein | 6-weeks
Pittsburgh Sleep Quality Index | 6-weeks
  The Pittsburgh Sleep Quality index, is a questionnaire that consists of 19 self-rated questions, grouped into 7 components. Each component is scored separately, weighted equally on a 0 - 3 scale and the scores of the 7 components are then added to give a global score, which has a range of 0 - 21 with higher scores indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Lancashire, Preston, Lancs, United Kingdom

IPD SHARING:
Plan to Share IPD: No